CLINICAL TRIAL: NCT04698642
Title: A 2-stage, Phase 1/2a Study to Evaluate the Safety, Tolerability, and Preliminary Efficacy of CBL-514 Injection for Reducing Convexity or Fullness of Abdominal Subcutaneous Fat (Phase 2a)
Brief Title: A Study to Evaluate the Safety, Tolerability, and Preliminary Efficacy of CBL-514 Injection for Reducing Convexity or Fullness of Abdominal Subcutaneous Fat
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Caliway Biopharmaceuticals Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CBL-16001(Phase 2a)
Record Dates: First submitted 2020-12-29; First posted 2021-01-07 (Actual); Last update posted 2021-01-08 (Actual); Status verified 2021-01

CONDITIONS: Subcutaneous Fat

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- CBL-514 180 mg, 1.2 mg/cm^2 (Experimental): CBL-514 will be administrated with the grid spacing of 2.5 cm^2
  Interventions: Drug: CBL-514
- CBL-514 240 mg, 1.6 mg/cm^2 (Experimental): CBL-514 will be administrated with the grid spacing of 2.5 cm^2
  Interventions: Drug: CBL-514
- CBL-514 300 mg, 2 mg/cm^2 (Experimental): CBL-514 will be administrated with the grid spacing of 2.5 cm^2
  Interventions: Drug: CBL-514

INTERVENTIONS:
Drug: CBL-514 — Both sides of the abdominal region will receive CBL-514.

SUMMARY:
The Phase 2a component of the study will be a randomized, open-label, parallel, and multiple dose study to further examine the safety and efficacy profile of 3 CBL-514 dose levels based on the results from Phase 1 of the study.

ELIGIBILITY:
Inclusion Criteria:

1. Male/female aged 18 years to 64 years old (at Screening), inclusive.
2. Body mass index >18.5 and <35 kg/m2 and body weight ≥50 kg at Screening and Day 1.
3. Has WC between 80.0 cm and 110.0 cm at Screening and Day 1.
4. Subcutaneous fat thickness of at least 3.00 cm (30.0 mm) and up to 6.00 cm (60.0 mm) by pinch method (measured by calibrated caliper) surrounding the center of treatment area at Screening and Day 1.
5. Subject has stable body weight for at least 3 months before Screening and during the study.
6. Subject who has maintained a stable lifestyle (e.g. exercise, eating patterns, and smoking habit) for at least 3 months before Screening and during the study.
7. Voluntarily signs the Informed Consent Form and, in the opinion of the Investigator or delegate, is physically and mentally capable of participating in the study, and willing to adhere to study procedures.

Exclusion Criteria:

1. Female subject of childbearing potential who is not willing to commit to an acceptable contraceptive regimen with her partner from the time of Screening and throughout study participation until 12 weeks after the last study drug dose, or who is currently pregnant or lactating. Male subject who is not willing to commit to an acceptable contraceptive method. For details on contraception, refer section 6.11.

   Females who have been surgically sterilized (hysterectomy or bilateral oophorectomy) or who are postmenopausal (e.g., defined as at least 50 years with ≥12 months of amenorrhea with a follicle stimulating hormone >40 IU/L) are considered to be of non-childbearing potential. Subjects who are not of childbearing potential are not required to use contraception.
2. Subject diagnosed with coagulation disorders or is receiving anticoagulant/antiplatelet therapy or medications or dietary supplements, which impede coagulation or platelet aggregation.
3. Subject has diabetes or glycated hemoglobin ≥6.5% (48 mmol/mol) or fasting blood sugar ≥7 mmol/L.
4. Subject has a clinically significant cardiovascular disease and abnormal findings in ECG.
5. Subject with active or prior history of malignancies (except for successfully treated basal cell carcinoma) within 5 years before Screening or being worked-up for a possible malignancy.
6. Subject with a history of human immunodeficiency virus (HIV)-1, hepatitis B, or hepatitis C infections or subjects with active HIV, hepatitis B, or hepatitis C infections at Screening:

   1. Active HIV infection: positive HIV Ag/Ab combo test;
   2. Active hepatitis B virus (HBV) infection: positive HBV surface antigen (HBsAg). Subjects with negative HBsAg but with positive HBV core antibody, with or without positive HBV surface antibody will also be excluded. However, subjects with negative HBsAg, negative HBV core antibody, and positive HBV surface antibody may be included.
   3. Active hepatitis C virus (HCV) infection: positive HCV antibody.
7. Subject has abnormal skin or local skin conditions at the treatment area, which in the opinion of Investigator is inappropriate to participate in the study, including but not limited to any of the following:

   1. Skin manifestations of a systemic disease,
   2. Any abnormality of the skin or soft tissues of the abdominal wall in the area to be treated,
   3. Skin or superficial tissue that does not lie flat on its own when the subject is in the supine position,
   4. Sensory loss or dysesthesia in the area to be treated,
   5. Evidence of any cause of enlargement in the abdominal area other than localized subcutaneous fat,
   6. Tattoos on the area to be treated.
8. Subject who has hernia
9. Subject who has undergone the following procedures:

   1. Previous open or laparoscopic abdominal surgery in the anticipated treatment area,
   2. Cardiac pacemakers or any implantable electrical device,
   3. Metal implants of any type in the area to be treated,
   4. Esthetic procedure i.e. liposuction to the region to be treated within 12 months before Screening or during the study,
   5. Esthetic procedure i.e. cryolipolysis, ultrasonic lipolysis, low level laser therapy , lipolysis injection to the region to be treated within 6 months before Screening or during the study.
10. Subject is on prescription or over-the-counter weight reduction medication or weight reduction programs within 3 months before Screening or during the study.
11. Subject is undergoing chronic steroid or immunosuppressive therapy.
12. Requiring continual use of the following therapeutic agents during the study:1 S-mephenytoin (Mesantoin), terfenadine (Teldane), buspirone (Buspar), fexofenadine (Fexotabs, Tefodine, Telfast, Xergic, Allegra).

    If a subject needs to use the above mentioned therapeutic agents during the study for any reason, these therapeutic agents should not be used at least for 2 days prior to dosing until 1 day post-dose, whichever is later.
13. Unable to receive topical anesthesia (e.g., history of hypersensitivity to lidocaine).
14. Subjects with known allergies or sensitivities to the study drug and/or excipients
15. Subjects with inadequate liver function at Screening defined as aspartate aminotransferase, alanine aminotransferase, alkaline phosphatase, total bilirubin, or gamma-glutamyl transferase >3.0 × ULN.
16. Subjects with inadequate renal function, defined as abnormal serum creatinine, and urea >1.5 × ULN or estimated glomerular filtration rate (eGFR) <60 mL/min/1.73 m2. Subjects who are currently on dialysis should be excluded.
17. Use of other investigational drug or device within 4 weeks prior to Screening.

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 43 (Actual)
Dates: Start 2020-02-03 (Actual); Primary Completion 2020-11-12 (Actual); Study Completion 2020-11-12 (Actual)

PRIMARY OUTCOMES:
Change of abdominal subcutaneous fat volume | Up to 8 weeks after last treatment
  Change of abdominal subcutaneous fat volume as measured by ultrasound around the treated area compared to Baseline

SECONDARY OUTCOMES:
Change of abdominal subcutaneous fat thickness | Up to 8 weeks after last treatment
  Change of abdominal subcutaneous fat thickness as measured by ultrasound-determined subcutaneous fat thickness over the treated area compared to Baseline,
Incidence of treatment emergent adverse events (TEAEs) | Up to 8 weeks after last treatment
  Number of participants experiencing TEAEs and number of individual TEAEs among treatment groups by severity and relationship to investigational product (IP)
Number of participants with clinically significant abnormalities in clinical laboratory values | Up to 4 weeks after last treatment
  Clinical laboratory tests include Biochemistry, Hematology, Coagulation and Urinalysis test
Number of participants with clinically significant abnormalities in vital signs | Up to 8 weeks after last treatment
  Vital signs measurements include temperature, pulse rate, blood pressure, and respiratory rate
Number of participants with clinically significant abnormalities in Electrocardiogram (ECG) | Up to 4 weeks after last treatment
  ECG parameters include heart rate, RR interval, PR interval, QT interval, QTc interval, and QRS interval
Number of participants with clinically significant abnormalities in physical examination | Up to 8 weeks after last treatment
  Physical examinations include assessment of cardiovascular, respiratory, gastrointestinal, and neurological systems
Number of participants with injection site reactions | Up to 8 weeks after last treatment
  Injection site reactions include but not limited to redness, swelling, bruising, tenderness, itching, pain, warmth, discoloration and hardness

CONTACTS AND LOCATIONS:
Locations (1):
- Investigational site, Melbourne, Australia

IPD SHARING:
Plan to Share IPD: No